CLINICAL TRIAL: NCT03800654
Title: Mindful Action for Pain: An Integrated Approach to Improve Chronic Pain Function
Brief Title: Mindful Action for Pain
Acronym: MAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2807-W; RX002807 (Other Grant/Funding Number: VA RR&D)
Record Dates: First submitted 2019-01-08; First posted 2019-01-11 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Psychological Flexibility; Mindfulness Meditation
MeSH Terms: conditions — Chronic Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Group Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindful Action for Pain (MAP) Development (Other): In the first arm, MAP will be fully developed.
  Interventions: Behavioral: Mindful Action for Pain
- MAP vs. CBT-CP (Active Comparator): In the second arm, MAP will be compared to CBT-CP to establish feasibility of a larger, future trial.
  Interventions: Behavioral: Mindful Action for Pain; Behavioral: Cognitive Behavioral Therapy for Chronic Pain

INTERVENTIONS:
Behavioral: Mindful Action for Pain — MAP integrates formal mindfulness meditation with methods from Acceptance and Commitment Therapy and Dialectical Behavior Therapy.
  Other Names: MAP
Behavioral: Cognitive Behavioral Therapy for Chronic Pain — CBT-CP is the current gold standard psychosocial intervention for chronic pain and will be compared to MAP in the second arm of the study.
  Other Names: CBT-CP
  Arms: MAP vs. CBT-CP

SUMMARY:
An emerging scientific model that has been applied to chronic pain is the psychological flexibility (PF) model. PF refers to the ability to behave consistently with one's values even in the face of unwanted thoughts, feelings, and bodily sensations such as pain. Acceptance and Commitment Therapy (ACT) is the best known treatment derived from the PF model and is as effective as the gold standard Cognitive Behavioral Therapy (CBT), but falls short on achieving meaningful changes in functional improvement. Although ACT was designed to impact PF, methods from different treatment approaches are also consistent with the model. An experiential strategy that holds promise for enhancing PF is formal mindfulness meditation, a practice used to train non-judgmental awareness and attention to present-moment experiences, which has never been tested within the PF model. There is compelling theoretical and empirical rationale that the mechanisms underlying formal mindfulness meditation will bolster PF processes and thereby can be applied to facilitate functional improvement. To test this, the principal investigator, has developed a novel 8-week group-based intervention, Mindful Action for Pain (MAP), which integrates formal mindfulness meditation with experiential methods from different evidence-based treatment approaches in accordance with the PF model. MAP is designed such that daily mindfulness meditation practice is used to develop the capacity to more completely utilize strategies to address the key psychosocial barriers (e.g., pain catastrophizing) to optimal functioning.

This career development award (CDA-2) project consists of two phases. Phase 1 (years 1 - 2) consists of using qualitative and quantitative methods to iteratively develop and refine MAP over the course of 4 MAP cycles (n = 20). Phase 2 (years 3 - 5) consists of a pilot randomized controlled trial (RCT) (n = 86) of MAP vs. cognitive behavioral therapy (CBT) for chronic pain (CBT-CP) in order to establish feasibility of a future large-scale trial and estimate the preliminary impact of MAP. Functional improvement will be measured by reductions in pain interference (primary clinical outcome). Further, meditation adherence will be assessed to explore dose-response relationships with functional improvement, and objective measures of physical activity (actigraphy) will be captured to explore the psychophysical impact of MAP.

DETAILED DESCRIPTION:
Chronic pain, defined as persistent or episodic pain that does not resolve with treatment, affects up to 50% of Veterans, costs the nation between $560 and $635 billion dollars annually, and is associated with high rates of disability and low quality of life. According to the Veterans Health Administration (VHA), the goal of pain treatment is to improve physical and psychosocial functioning, emphasizing non-pharmacological approaches, such as psychosocial interventions, to target psychosocial factors that maintain disability. Unfortunately, the gold standard psychosocial intervention for chronic pain, Cognitive Behavioral Therapy (CBT), does not reliably produce meaningful increases in function.

An emerging scientific model that has been applied to chronic pain is the psychological flexibility (PF) model. PF refers to the ability to behave consistently with one's values even in the face of unwanted thoughts, feelings, and bodily sensations such as pain. Acceptance and Commitment Therapy (ACT) is the best known treatment derived from the PF model and is as effective as the gold standard CBT, but still falls short on achieving meaningful changes in functional improvement. Although ACT was designed to impact PF, methods from different treatment approaches are also consistent with the model. An experiential strategy that holds promise for enhancing PF is formal mindfulness meditation, a practice used to train non-judgmental awareness and attention to present-moment experiences, which has never been tested within the PF model. There is compelling theoretical and empirical rationale that the mechanisms underlying formal mindfulness meditation will bolster PF processes and thereby can be applied to facilitate functional improvement. To test this, the principal investigator, has developed a novel 8-week group-based intervention, Mindful Action for Pain (MAP), which integrates formal mindfulness meditation with experiential methods from different evidence-based treatment approaches in accordance with the PF model. MAP is designed such that daily mindfulness meditation practice is used to develop the capacity to more completely utilize strategies to address the key psychosocial barriers (e.g., pain catastrophizing) to optimal functioning.

This CDA-2 project consists of two phases. Phase 1 (years 1 - 2) consists of using qualitative and quantitative methods to iteratively develop and refine MAP over the course of 4 MAP cycles (n = 20). Phase 2 (years 3 - 5) consists of a pilot RCT (n = 86) of MAP vs. CBT for chronic pain (CBT-CP) in order to establish feasibility of a future large-scale trial and estimate the preliminary impact of MAP. Functional improvement will be measured by reductions in pain interference (primary clinical outcome). Further, meditation adherence will be assessed to explore dose-response relationships with functional improvement, and objective measures of physical activity (actigraphy) will be captured to explore the psychophysical impact of MAP.

Aim 1: Fully develop MAP in a population of Veterans with chronic pain (Phase 1).

Aim 2: Evaluate the feasibility of a future randomized efficacy trial of MAP vs. CBT-CP (Phase 2).

Hypothesis 1: MAP and CBT-CP will be feasible to deliver, as evidenced by attainment of recruitment goals, retention rates > 80%, and high credibility and expectancy ratings.

Aim 3: Estimate the preliminary impact of MAP and CBT-CP to determine if a future efficacy trial is warranted.

Examine changes in pain interference (a proxy for functional improvement and one of the most commonly measured outcomes in psychosocial intervention trials of chronic pain), pain acceptance, trait mindfulness, and pain catastrophizing, as well as patient satisfaction ratings, as indicators that MAP may be worthy of investigation in a future large-scale trial.

Exploratory Aim 1: Explore the relationship between meditation adherence and treatment outcomes.

There is growing evidence for a dose-response relationship between meditation practice and positive outcomes. Therefore, strategies to increase meditation adherence will be optimized (Phase 1) and the relationship between adherence as measured via daily diaries and outcomes will be assessed (Phase 2).

Exploratory Aim 2: Explore objective measures of physical activity at baseline and post-intervention as a potential future index of functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Diagnosis of a chronic, non-terminal pain condition
* Pain most days (> 3 days/week) for at least 6 months
* Average pain severity and interference with enjoyment of life and/or general activity rated > 4/10 over the past week

Exclusion Criteria:

* Serious or unstable medical or psychiatric illness

  * (e.g., unmanaged psychosis, manic episode, or substance abuse within the past year) or psychosocial instability
  * (e.g., homelessness) that could compromise study participation
* Active suicidal ideation or history of suicide attempt within past 3 years
* Current participation in group psychotherapy for pain or any type of individual psychotherapy
* Changes to professionally delivered pain or mood treatments

  * (e.g., no discontinuation of a treatment; no increasing the dose of medication) one month preceding the baseline assessment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2024-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Herbert, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
A data repository will be created upon completion of the study. Data obtained in this study that has scientific value to other qualified researchers will made available upon request. Interested researches will be able to access de-identified data through a Data Use Agreement.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Indefinitely
Access Criteria: February, 2024

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 126 participants completed the informed consent procedure. However, 9 of these participants either declined or were excluded prior to assigning them to an intervention and 1 participant did not complete the baseline assessment (violating are intent-to-treat criterion). Thus, only 116 (Phase 1: n=29; Phase 2: n=87) were assigned to an intervention and completed the baseline assessment.
Groups:
- Mindful Action for Pain (MAP) Development (Years 1-2): In the first arm, MAP will be fully developed.
  Mindful Action for Pain: MAP integrates formal mindfulness meditation with methods from Acceptance and Commitment Therapy and Dialectical Behavior Therapy.
- MAP (Years 3-5): Mindful Action for Pain: MAP integrates formal mindfulness meditation with methods from Acceptance and Commitment Therapy and Dialectical Behavior Therapy.
- CBT (Years 3-5): Cognitive Behavioral Therapy for Chronic Pain: CBT-CP is the current gold standard psychosocial intervention for chronic pain and will be compared to MAP in the second arm of the study.
Period: Overall Study
Arm/Group | Mindful Action for Pain (MAP) Development (Years 1-2) | MAP (Years 3-5) | CBT (Years 3-5)
Started | 29 | 46 | 41
Completed | 23 | 39 | 31
Not Completed | 6 | 7 | 10
Not completed — Time constraints | 3 | 3 | 3
Not completed — Did Not Meet Inclusion Criteria | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 6
Not completed — Medical Health Issue | 0 | 0 | 1
Not completed — Personal Issues | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mindful Action for Pain (MAP) Development (Years 1-2): In the first arm, MAP will be fully developed.
  Mindful Action for Pain: MAP integrates formal mindfulness meditation with methods from Acceptance and Commitment Therapy .
- MAP (Years 3-5): Mindful Action for Pain: MAP integrates formal mindfulness meditation with methods from Acceptance and Commitment Therapy .
- Total: Total of all reporting groups
Arm/Group | Mindful Action for Pain (MAP) Development (Years 1-2) | MAP (Years 3-5) | CBT (Years 3-5) | Total
Number analyzed (Participants) | 29 | 46 | 41 | 116
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: 2 phases of project
  Years | 57.28 (13.92) | 50.83 (12.21) | 47.88 (12.62) | 51.40 (13.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 10 | 26
  Male | 23 | 36 | 31 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 10 | 10 | 27
  Not Hispanic or Latino | 22 | 35 | 31 | 88
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 1 | 5 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 8 | 13 | 13 | 34
  White | 9 | 18 | 18 | 45
  More than one race | 1 | 3 | 1 | 5
  Unknown or Not Reported | 10 | 6 | 4 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 46 | 41 | 116
Brief Pain Inventory - Pain Interference [Mean (Standard Deviation); unit: units on a scale] — The BPI Pain Interference subscale consists of 7-items rated on a 0 - 10 scale that measures the degree to which pain interferes with various aspects of life, including mobility, social activities, and mood. Scores are averaged with a range from 0 to 10. Higher scores indicate higher levels of pain interference (i.e., worse outcome).
  units on a scale | 6.77 (1.66) | 7.31 (1.76) | 7.38 (1.95) | 7.20 (1.81)

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory (BPI) Pain Interference Subscale Change
Description: The BPI Pain Interference subscale consists of 7-items rated on a 0 - 10 scale that measures the degree to which pain interferes with various aspects of life, including mobility, social activities, and mood. Scores are averaged with a range from 0 to 10. Higher scores indicate higher levels of pain interference (i.e., worse outcome).
Time Frame: Baseline and week 9
Population: Veterans with heterogenous chronic pain
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mindful Action for Pain (MAP) Development (Years 1-2): In the first arm, MAP will be fully developed.
  Mindful Action for Pain: MAP integrates formal mindfulness meditation with methods from Acceptance and Commitment Therapy.
- MAP Group (Years 3-5): In Years 3-5, MAP will be compared to CBT-CP to establish feasibility of a larger, future trial.
  Mindful Action for Pain: MAP integrates formal mindfulness meditation with methods from Acceptance and Commitment Therapy.
- CBT Group (Years 3-5): In Years 3-5, MAP will be compared to CBT-CP to establish feasibility of a larger, future trial.
  Cognitive Behavioral Therapy for Chronic Pain: CBT-CP is the current gold standard psychosocial intervention for chronic pain and will be compared to MAP in the second arm of the study.
Arm/Group | Mindful Action for Pain (MAP) Development (Years 1-2) | MAP Group (Years 3-5) | CBT Group (Years 3-5)
Number analyzed (Participants) | 29 | 46 | 41
units on a scale
  Baseline | 6.77 (1.66) | 7.31 (1.76) | 7.38 (1.95)
  Post-treatment: number analyzed (Participants) | 29 | 39 | 31
  Post-treatment | 5.40 (2.32) | 6.19 (2.04) | 5.63 (2.20)

2. Secondary Outcome: Chronic Pain Acceptance Questionnaire (CPAQ)
Description: The CPAQ consists of 20-items rated on a 0 - 6 scale that measures the degree that patients have adjusted to pain as part of their identity and lifestyle. Scores range from 0 to 120. Higher scores indicate higher levels of pain acceptance (i.e., better outcome).
Time Frame: Baseline and week 9
Population: Veterans with heterogenous chronic pain
Measure: Mean (Standard Deviation); unit: units on scale
Groups:
- MAP (Years 3-5): Mindful Action for Pain: MAP integrates formal mindfulness meditation with methods from Acceptance and Commitment Therapy.
Arm/Group | Mindful Action for Pain (MAP) Development (Years 1-2) | MAP (Years 3-5) | CBT (Years 3-5)
Number analyzed (Participants) | 29 | 46 | 41
units on scale
  Baseline | 65.55 (11.54) | 63.50 (10.80) | 62.78 (9.72)
  Posttreatment: number analyzed (Participants) | 29 | 39 | 31
  Posttreatment | 72.78 (7.90) | 65.23 (14.02) | 67.03 (8.99)

3. Secondary Outcome: Mindfulness Attention Awareness Scale (MAAS)
Description: The MAAS consists of 15-items assessing present-moment attention and awareness of everyday experiences. Scores range from 1-6 with higher scores reflecting greater mindfulness (i.e., better outcome).
Time Frame: Baseline and week 9
Population: Veterans with heterogenous chronic pain
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Mindful Action for Pain (MAP) Development (Years 1-2) | MAP (Years 3-5) | CBT (Years 3-5)
Number analyzed (Participants) | 29 | 46 | 41
units on scale
  Baseline | 3.62 (1.00) | 3.87 (1.07) | 3.55 (1.00)
  Posttreatment: number analyzed (Participants) | 29 | 39 | 31
  Posttreatment | 3.93 (.80) | 3.97 (1.01) | 3.63 (1.18)

4. Secondary Outcome: Pain Catastrophizing Scale (PCS)
Description: The PCS consists of 13 items rated on 0 - 4 scale that measures the degree to which people experience an aversive orientation towards pain. Scores range from 0 - 52). Higher scores indicate higher levels of pain catastrophizing (i.e., worse outcome).
Time Frame: Baseline and week 9
Population: Veterans with heterogenous chronic pain
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Mindful Action for Pain (MAP) Development (Years 1-2) | MAP (Years 3-5) | CBT (Years 3-5)
Number analyzed (Participants) | 28 | 45 | 41
units on scale
  Baseline | 26.86 (12.29) | 28.98 (11.31) | 27.80 (12.25)
  Posttreatment: number analyzed (Participants) | 28 | 39 | 31
  Posttreatment | 21.74 (10.66) | 22.72 (11.88) | 21.52 (12.49)

5. Other Pre Specified Outcome: Meditation Diaries
Description: On these diaries, participants report the duration of meditation practice and what kind of practice (e.g., breathing, body scan).
Time Frame: Weekly during treatment (i.e., weeks 1 - 8) and week 9
Reporting Status: Not Posted, anticipated posting 2025-11

6. Other Pre Specified Outcome: Actigraphy
Description: Participants will wear actiwatches for two 7-day periods at baseline and week 9 to measure average physical activity counts.
Time Frame: Baseline and week 9
Reporting Status: Not Posted, anticipated posting 2025-11

ADVERSE EVENTS:
Time Frame: Baseline through study completion, an average of 3 months post-treatment
Description: Does not differ
Arm/Group | Mindful Action for Pain (MAP) Development (Years 1-2) | MAP (Years 3-5) | CBT (Years 3-5)
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/46 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/46 | 0/41
Other Adverse Events (participants affected / at risk) | 0/29 | 0/46 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT03800654/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT03800654/ICF_001.pdf